CLINICAL TRIAL: NCT05579756
Title: Psychatric Impact of Miscarriage and Its Associated Factors Among Women in Assiut University Women's Health Hospital
Brief Title: Psychatric Impact of Miscarriage in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mostafa, Dr, Assiut University
Other Study IDs: miscarriag
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Miscarriage is basically defined as intrauterine fetal death before viability (1,2). Age of viability, in Egypt, sets at 26 weeks of gestation (3). Incidence of miscarriage is often referred to as an iceberg where the actual size of the problem cannot be determined. More than 50% of human conceptions are lost before the missed period either before or after implantation (4). In clinically recognized pregnancies, losses decrease as pregnancy progresses from 17% - 20 % after 6 weeks to only 3% at 10 weeks gestation (4). Beside the high incidence of miscarriage, it implies a high psychological morbidity to both partners with increased liability to anxiety, post stress disorder and depression(5,6). This psychological impact can be attributed not only to loss of desired child but also to the traumatic event of bleeding and pain encountered by those patients (7).

DETAILED DESCRIPTION:
Miscarriage is basically defined as intrauterine fetal death before viability (1,2). Age of viability, in Egypt, sets at 26 weeks of gestation (3). Incidence of miscarriage is often referred to as an iceberg where the actual size of the problem cannot be determined. More than 50% of human conceptions are lost before the missed period either before or after implantation (4). In clinically recognized pregnancies, losses decrease as pregnancy progresses from 17% - 20 % after 6 weeks to only 3% at 10 weeks gestation (4). Beside the high incidence of miscarriage, it implies a high psychological morbidity to both partners with increased liability to anxiety, post stress disorder and depression(5,6). This psychological impact can be attributed not only to loss of desired child but also to the traumatic event of bleeding and pain encountered by those patients (7).

While the clinical management of miscarriage and its physical complications have been extensively discussed; the psychological impact of this traumatic event of loss is usually overlooked especially in developing countries (8-11). Moreover, there are behind-the-scene factors that trigger or correlate to the development of psychiatric morbidities following miscarriage (12,13). Factors as sociodemographic, marital satisfaction, social support, individual's coping resources, history of infertility and previous miscarriage vary across different population samples, also vary in their influence on women's psychological resilience after traumatic events as miscarriage. No previous studies addressed this topic in Egyptian population.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women 18:45 years old presented by intrauterine pregnancy loss before <= 26 weeks gestation

Exclusion Criteria:

* Ectopic pregnancy or vesicular mole
* previous diagnosis of psychatric disorder
* unwell to give consent

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: - all pregnant women 18:45 years old presented by intrauterine pregnancy loss before <= 26 weeks gestation
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
prevelance of post traumatic stress disorder , depression, and anxiety one month after miscarriage | 1 year maximum